CLINICAL TRIAL: NCT02712970
Title: A Proposed Staging System for Chronic Symptomatic Pilonidal Sinus Disease and Results in Patients Treated With Stage-based Approach
Brief Title: Staging System for Chronic Symptomatic Pilonidal Sinus Disease
Status: Completed | Type: Observational
Sponsor: Trabzon Numune Training and Research Hospital (Other Government)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali GUNER, MD, MD, Trabzon Numune Training and Research Hospital
Other Study IDs: TrabzonNTRH
Record Dates: First submitted 2016-03-05; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- stage-I: Single pit in the midline, no lateral extension. Pit-picking technique will be performed.
  Interventions: Procedure: pit-picking technique
- Stage-II: >1 pits in the midline, no lateral extension. Pit-picking and Bascom cleft lift techniques will be performed.
  Interventions: Procedure: pit-picking technique; Procedure: Bascom Cleft Lift
- Stage-III: Midline pit/pits plus lateral extension in one direction. Bascom cleft lift technique will be performed.
  Interventions: Procedure: Bascom Cleft Lift
- Stage-IV: Midline pit/pits plus lateral extension in both directions. Rhomboid excision with the Limberg Flap will be performed.
  Interventions: Procedure: Rhomboid excision with the Limberg Flap
- Stage-R: Recurrent PSD following any type of treatment. Other flap techniques such as V-Y advancement flap, Z-Plasty will be performed.
  Interventions: Procedure: Bascom Cleft Lift; Procedure: Rhomboid excision with the Limberg Flap; Procedure: Other flap techniques

INTERVENTIONS:
Procedure: pit-picking technique — midline pits were excised removing a minimal amount of tissue (with a margin of skin of <1 mm). Incision of 1-2 cm in length was performed parallel to the most convenient side of the midline to be curetted of the chronic abscess cavity. All infected granulation tissue and hair were removed. After establishing hemostasis, the area of the excised midline pits was approximated by absorbable sutures.
  Groups: Stage-II; stage-I
Procedure: Bascom Cleft Lift — The upper end of the incision was made 1-2 cm lateral to the midline on the more affected side and this was continued vertically over a distance of 1-2 mm from the midline pits. The lower end was fashioned from the midline in a V-shape in order to prevent a dog-ear deformity. The skin on this side of the natal cleft was then elevated and excised. The skin on the opposite side was undermined to the distance required to allow primary closure of the defect away from the midline without tension. Sinus tissue and its extensions were excised. The incision was then closed subcuticularly by absorbable polyglecaprone (3-0), after which a few interrupted mattress polyglecaprone (3-0) buttress sutures were also inserted.
  Groups: Stage-II; Stage-III; Stage-R
Procedure: Rhomboid excision with the Limberg Flap — The area to be excised was mapped on the skin in a rhomboid form, and the flap was designed. The skin incision was deepened to the postsacral fascia. The flap was fully mobilized and transposed medially to fill the defect without tension. The wound was closed in two layers: the subcutaneous tissue with absorbable (2/0 polyglactin) sutures and the skin with nonabsorbable (3/0 polypropylene) interrupted mattress suture
  Groups: Stage-IV; Stage-R
Procedure: Other flap techniques — Bascom Cleft lift as described above, Rhomboid excision with the Limberg Flap as described above, V-Y advancement flap, Z-Plasty
  Groups: Stage-R

SUMMARY:
A staging system was defined based on morphological extent of disease (stage I to stage IV for primary disease, and stage R for recurrent disease). Specific surgical technique was used for each stage. Demographics, perioperative data, short-term and long-term outcomes were evaluated according to the disease stage.

DETAILED DESCRIPTION:
The collected data of patients who underwent surgery for the treatment of pilonidal sinus disease prior to June 2011 were analyzed. Following this analysis, a staging system was defined based on morphological extent of disease (stage I to stage IV for primary disease, and stage R for recurrent disease). Specific surgical technique was used for each stage. "Pit-picking" technique was performed under local anesthesia on an outpatient basis in stage I and stage IIa patients. For stage IIb and stage III patients, the Bascom Cleft Lift /modified Bascom Cleft Lift techniques were performed. For stage IV patients, the rhomboid excision with the Limberg flap technique was used. Demographics, perioperative data, short-term and long-term outcomes were evaluated according to the disease stage.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with symptomatic pilonidal sinus disease.

Exclusion Criteria:

* <18 y
* Pilonidal sinus disease which identified incidentally and which presented with acute abscesses were not included to the staging system.
* Patients who were treated without the use of the suggested algorithm were excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were operated because of chronic symptomatic pilonidal sinus disease
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Early wound complications | up to 3 months
  Complications were classified as infection (superficial or deep), collection (seroma or hematoma), wound dehiscence (partial or complete), or anesthesia-related complications. complications will be reviewed from time of surgery to the end of healing. percentage of participants with any wound complication will be evaluated as patients with complication.

SECONDARY OUTCOMES:
Assessment of recurrence (recurrence is defined when symptoms of the disease recurred after an interval following complete wound healing.) | 3 years
  Patients will be followed up for recurrence for three years. Total number of patients presenting with recurrence will be evaluated at the end of 3rd year.
Primary healing rate | within 3 months
  All surgical site complications were recorded, and patients with prolonged healing were regularly examined until complete healing was achieved. Primary healing was defined as no breakdown of the wound (complication-free healing) at any point along its length.
Hospital stay "The interval from the day of surgery to the day of discharge was recorded as the ''hospital stay.'' | during first week (one week)
  hospital stay for patients in postoperative period will be measured from the day of surgery to the day of discharge (as days).
Operative duration (''Operative duration'' is defined as the time between the initiation of the incision and the application of the last suture.) | during surgery

IPD SHARING:
Plan to Share IPD: No
because this is retrospective study.

REFERENCES:
- [Background] Guner A, Boz A, Ozkan OF, Ileli O, Kece C, Reis E. Limberg flap versus Bascom cleft lift techniques for sacrococcygeal pilonidal sinus: prospective, randomized trial. World J Surg. 2013 Sep;37(9):2074-80. doi: 10.1007/s00268-013-2111-9. PMID 23732258
- [Background] Guner A, Ozkan OF, Kece C, Kesici S, Kucuktulu U. Modification of the Bascom cleft lift procedure for chronic pilonidal sinus: results in 141 patients. Colorectal Dis. 2013 Jul;15(7):e402-6. doi: 10.1111/codi.12243. PMID 23581906
- [Background] Bascom J, Bascom T. Utility of the cleft lift procedure in refractory pilonidal disease. Am J Surg. 2007 May;193(5):606-9; discussion 609. doi: 10.1016/j.amjsurg.2007.01.008. PMID 17434365
- [Background] Mentes O, Bagci M, Bilgin T, Ozgul O, Ozdemir M. Limberg flap procedure for pilonidal sinus disease: results of 353 patients. Langenbecks Arch Surg. 2008 Mar;393(2):185-9. doi: 10.1007/s00423-007-0227-9. Epub 2007 Sep 22. PMID 17899165
- [Background] Can MF, Sevinc MM, Hancerliogullari O, Yilmaz M, Yagci G. Multicenter prospective randomized trial comparing modified Limberg flap transposition and Karydakis flap reconstruction in patients with sacrococcygeal pilonidal disease. Am J Surg. 2010 Sep;200(3):318-27. doi: 10.1016/j.amjsurg.2009.08.042. Epub 2010 Feb 1. PMID 20122682
- [Background] Kement M, Oncel M, Kurt N, Kaptanoglu L. Sinus excision for the treatment of limited chronic pilonidal disease: results after a medium-term follow-up. Dis Colon Rectum. 2006 Nov;49(11):1758-62. doi: 10.1007/s10350-006-0676-1. PMID 16990977
- [Derived] Guner A, Cekic AB, Boz A, Turkyilmaz S, Kucuktulu U. A proposed staging system for chronic symptomatic pilonidal sinus disease and results in patients treated with stage-based approach. BMC Surg. 2016 Apr 16;16:18. doi: 10.1186/s12893-016-0134-5. PMID 27084534